CLINICAL TRIAL: NCT06302127
Title: County Medical Community-based, Cardiovascular Risk Stratified Integrated Care Model: a Pragmatic Cluster Randomised Control Trial
Acronym: C-RISIMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CCHDS
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hypertension; Diabetes Mellitus Type 2; Cardiovascular Diseases
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The follow-up data collection, data entry, and data quality checks will be conducted by researchers unaware of the group assignments. The analysis of results will also be performed by statisticians unaware of the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): During the study, control participant will be provided with existing essential public health service including quarterly follow-ups and annual physical examination, and be advised to see their usual provider for care, as appropriate.
- Intervention (Experimental): Intervention group will receive the risk-stratified integrated CVD management (RISIMA) model consisting of 5 core elements provided as a package: (1) Team-based care; (2) Risk-stratified care pathway; (3) Strengthened health education; (4) Financial incentives for integration of care; (5) Supporting health information system.
  Interventions: Other: Team-based care; Procedure: Risk-stratified care pathway; Behavioral: Strengthened health education; Other: Financial incentives for integration of care; Other: Supporting health information system

INTERVENTIONS:
Other: Team-based care — The RISIMA model is provided by a family healthcare team composed of one village doctor, one general physician at township health centers and one specialist including cardiologists, neurologists or endocrinologists from county hospital. For villages without village doctor, public health professionals from township health centers would join the service team as the supplement. Within the team, three team members carry the different function. Village doctor is responsible for regular home visits, CVD risk measurement and organizing health education course. GP as the core service provider in the team is responsible for CVD risk monitoring, providing health education course for middle-high risk participants, and generating integrated care plans for each participant. Specialist is responsible for providing guidance particularly for high-risk population management to township and village doctors within the team.
  Arms: Intervention
Procedure: Risk-stratified care pathway — Based on WHO/ISH score, baseline population will be divided into three groups-low risk (10-year CVD risk: <10%), middle risk (10-year CVD risk: 10%~20%) and high risk (10-year risk: >20%). With the support from experts and health care professionals, study had developed a risk-stratified care pathway on the basis of clinical guidance. According to the pathway, participants at different risk tertile are provided with differentiated management plan especially in terms of health education, follow-up frequency and treatment plan.
  Arms: Intervention
Behavioral: Strengthened health education — The education comprised 8 monthly sessions developed by GP and village doctors. At the 4th month, individual health counseling by village doctors will be done to encourage the imitation and maintenance of self-management behaviors, and to identify any potential problems in the program. It took half an hour per each participant. At the 8th month, self-management evaluation will be done to assess personal self-management ability. High risk participants are required to take the education course, and middle risk participants are only encouraging to take. All participants would receive the education messages twice a month, which introduce tips about the management of hypertension, diabetes and CVD risk factors.
  Arms: Intervention
Other: Financial incentives for integration of care — Specialists receive reimbursement for case discussion and high risk population management; GP receive reimbursement for providing education program and risk monitoring; Village doctor receive reimbursement for assisting education program, risk measurement and home visits. And overall services quality will be measured, and taken into account for annual performance evaluation.
  Arms: Intervention
Other: Supporting health information system — A dynamic patient risk monitoring information system is established for simplifying the risk data collection and entry for village doctors, meanwhile, GP and specialist can receive the updates of risk scores simultaneously. Apart from the function of risk monitoring, this system also incorporates the e-records of home visits, health education attendance as well as medical records including outpatient visits and hospitalizations. The upgraded information systems not only can support the healthcare professionals with comprehensive and real-time data, but also provide the performance evaluation data for policymakers.
  Arms: Intervention

SUMMARY:
The goal of this cluster randomized trial is to evaluate the effectiveness of the RISIMA model based on an integrated county healthcare consortium implemented by multi-level family health teams (FHTs)on patients with diabetes and/or hypertension, including CVD risk assessment, treatment, and management.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 40 and 70 years old;
2. Patients with hypertension or diabetes;
3. Permanent residents of the county where the research is conducted;
4. Already signed up with the family doctor team in the township where the research is located.

Exclusion Criteria:

1. Unable to independently carry out the interventions required for the study;
2. Residing far from the village or township health center where the research is located, making it difficult to cooperate with visits;
3. Patients who refuse to participate;
4. Patients with comorbidities such as cancer that may interfere with the study visits or intervention effects;
5. Pregnant or lactating women

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2560 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
10-year CVD risk score | 12 months
  This study intervention is designed to address CVD risk by introducing an integrated care package. Therefore, a validated risk score is required to properly evaluate the effect of interventions. The WHO/ISH score is a tool to estimate the risk of CVD development based on age, sex, BP, total cholesterol, smoking and diabetes. The primary objective of this study is to evaluate whether or not the intervention can substantially lower the risk at 1 year. The primary outcome is the mean difference in WHO/ISH risk score change from baseline to 12 months between the intervention and control townships. The WHO/ISH risk score will be calculated using the lab-based measurements, but if there are missing, a nonlaboratory measurements will be used.

SECONDARY OUTCOMES:
10-year CVD risk score changes | 6 months
  change in 10-year CVD risk score changes between the intervention and control FDTs at 6 months
blood pressure control rate | 12 months
  change in blood pressure control rate between the intervention and control FDTs at 12 months
systolic blood pressure | 12 months
  change in SBP between the intervention and control FHTs at 12 months
systolic blood pressure | 6 months
  change in SBP between the intervention and control FHTs at 6 months
total cholesterol | 12 months
  change in total cholesterol between the intervention and control FHTs at 12 months.
fasting blood glucose | 12 months
  change in fasting blood glucose between the intervention and control FDTs at 12 months
CVD incidence rate | 12 months
  difference of incidence rate of major adverse cardiovascular events (including acute myocardial infarction, stroke, angina, and sudden cardiac death) between the intervention and control FDTs at 12 months
cost-effectiveness outcome | 12 months
  a health economic evaluation to assess the cost-effectiveness of the intervention compared with usual care at 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Shaxian County General Hospital, Sanming, Fujian
  - Luzhai County People's hospital, Liuchow, Guangxi
  - Luzhai County Traditional Medicine hospital, Liuchow

IPD SHARING:
Plan to Share IPD: No